CLINICAL TRIAL: NCT01492894
Title: A Randomized Controlled Trial of Reducing Calcineruin Inhibitor Target Level by 50% Versus Converting to Rapamycin in Chronic Kidney Dysfunction Without Reversible Causes
Brief Title: Kidney Allograft Dysfunction Without Reversible Causes
Acronym: KADWORC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study terminated due to low enrollment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0708M13942
Record Dates: First submitted 2010-08-09; First posted 2011-12-15 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Kidney Graft Dysfunction
MeSH Terms: interventions — Cyclosporins; Tacrolimus; Cyclosporine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50% decrease in calcineurin inhibitor (Active Comparator)
  Interventions: Drug: Cyclosporins/Tacrolimus
- Rapamune (Active Comparator)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Cyclosporins/Tacrolimus — Decrease the dose of calcineurin inhibitor by 1/2 and the drug level will be followed and adjusted to the target level of 50% of the previous levels
  Other Names: Gengraf (cyclosporin); Neoral (cyclosporin); Prograf (tacrolimus)
  Arms: 50% decrease in calcineurin inhibitor
Drug: Sirolimus — Change from current calcineurin inhibitor to Sirolumus
  Other Names: Rapamune
  Arms: Rapamune

SUMMARY:
The purpose of this study is to learn the best way to prolong kidney life in patients exposed to calcineurin inhibitors, who already have evidence of damage possibly caused by the calcineurin inhibitor on kidney biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Serum creatinine increased greater than or equal to 25% over baseline with no acute or reversible cause clinically evident.

   Although eGFR is arguably better for estimating kidney allograft function than serum creatinine, pragmatics dictate the use of a change in serum creatinine in the initial selection of patients. These criteria are currently used by transplant coordinators for selection of patients for the kidney biopsy as a part of large on-going study at our center.
2. Adequate (greater than or equal to 8 glomeruli) biopsy showing Chronic allograft injury reported as mild/moderate CAN or CNI toxicity based on the previously used Banff 97 classification and no potentially reversible causes of graft dysfunction, e.g. acute rejection or treatable recurrent disease. Patients with histological evidence of mild recurrent disease that does not appear to be severe enough to explain the deterioration in function, e.g. IgA on immunofluorescence, or changes consistent with early diabetic nephropathy, will not be excluded.
3. Receiving CsA (trough level concentration 75-125 ng/mL) or Tacrolimus(trough level concentration 6-12 ng/mL) plus MMF (or AZA) with (or without) prednisone.
4. Able to give informed consent.

Exclusion Criteria:

1. Urine total protein excretion >500 mg/g creatinine.
2. eGFR (estimated by MDRD) <40 mL/min/1.73 m2
3. Triglycerides >400 mg/dL or total cholesterol >300 mg/dL
4. Allergy to macrolide antibiotic or rapamycin
5. Women of child-bearing potential not using effective contraception
6. Treated for acute rejection within the past 2 months
7. <12 months after transplantation
8. Potentially treatable cause(s) of allograft dysfunction, including acute rejection, dehydration, and congestive heart failure.
9. Recurrent or de novo kidney disease that is histologically severe enough to be causing graft dysfunction
10. Polyoma virus (BK) nephropathy, or serum positive for BK by polymerase chain reaction
11. A second, functioning organ transplant.
12. Receiving sirolimus.
13. Patients with any past or present malignancy (other than non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Kidney function will be determined by the rate of change in glomerular filtration rate (GFR), estimated by serum creatinine (eGFR). | Once a week for 3 month then monthly until trial ends

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Kukula, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Departments of Medicine and Surgery, Minneapolis, Minnesota, United States